CLINICAL TRIAL: NCT04525157
Title: A Two-Arm, Randomized, Double-Blind, Phase IIb Study to Compare the Efficacy and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants Plus Narrow-Band Ultraviolet B (NB-UVB) Light Source With Narrow-Band Ultraviolet B (NB-UVB) Light Source in the Treatment of Nonsegmental Vitiligo AND A Single-Arm, Open Label, Phase IIb Study to Evaluate the Efficacy and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants Plus Narrow-Band Ultraviolet B (NB-UVB) Light Source in the Treatment of Nonsegmental Vitiligo
Brief Title: Afamelanotide and Narrow-Band Ultraviolet B (NB-UVB) Phototherapy in the Treatment of Nonsegmental Vitiligo (NSV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CUV103
Record Dates: First submitted 2020-08-06; First posted 2020-08-25 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — afamelanotide

STUDY DESIGN:
Intervention Model Description: A Two-Arm, Randomized, Double-Blind Study and a Single-Arm, Open Label, Phase IIb Study to Evaluate the Efficacy and Safety of Subcutaneous, Bioresorbable Afamelanotide Implants plus Narrow-Band Ultraviolet B (NBUVB) Light Source in the Treatment of Nonsegmental Vitiligo.
Who Masked: Participant, Investigator
Masking Description: In the first half of the study, the Participant and Investigator are masked. In the second half of the study, the study is single arm, Open Label Study.

ARMS (3):
- Afamelanotide and NB-UVB (Experimental): Participants received Afamelanotide implants (Days 28, 56, 112, 140, and 168) and NB-UVB light (twice weekly for 7 months from Day 0).
  Interventions: Drug: Afamelanotide
- Placebo and NB-UVB (Placebo Comparator): Participants received Placebo implants (Days 28, 56, 112, 140, and 168) and NB-UVB light (twice weekly for 7 months from Day 0).
  Interventions: Drug: Placebo
- Single-Arm, Open Label Group (Experimental): The study design was modified into a single-arm, open label study with only one treatment group receiving afamelanotide implants plus NB-UVB light.
  Participants received Afamelanotide implants (Days 28, 56, 112, 140, and 168) and NB-UVB light (twice weekly for 7 months from Day 0).
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide
  Arms: Afamelanotide and NB-UVB; Single-Arm, Open Label Group
Drug: Placebo
  Arms: Placebo and NB-UVB

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of afamelanotide, when combined with narrowband ultraviolet B (NB-UVB) phototherapy, in patients with nonsegmental vitiligo. Afamelanotide is expected to increase the rate of the repigmentation induced by NB-UVB, leading to a reduced frequency and dose of NB-UVB.

DETAILED DESCRIPTION:
Vitiligo is the most common depigmentation disorder. A commonly used treatment is phototherapy with narrow-band ultraviolet B irradiation (NB-UVB). Further therapeutic approaches are desired and currently being evaluated. The investigational product, afamelanotide, is a synthetic analogue of the human alpha melanocyte stimulating hormone (alpha-MSH). Afamelanotide activates melanin in skin, with the controlled-release injectable implant formulation having an affect across the total body surface area (pandermally). Earlier studies in vitiligo patients showed afamelanotide, in combination with NB-UVB, could induce faster and deeper repigmentation in patients compared to NB-UVB alone.

ELIGIBILITY:
Inclusion Criteria:

* for double-blind phase: Male and female subjects with a confirmed diagnosis of nonsegmental vitiligo with 15% to 50% of total body surface involvement
* for open label phase: Male and female subjects with a confirmed diagnosis of nonsegmental vitiligo with 10% to 50% of total body surface involvement
* Vitiligo involving the head and neck
* Stable or slowly progressive vitiligo over a 3-month period
* Aged 21 years or more
* Willing and able to comply with the conditions specified in this protocol and study procedures, in the opinion of the Investigator
* Provided written Informed Consent prior to the performance of any study-specific procedure

Exclusion Criteria:

* Extensive leukotrichia, in the opinion of the Investigator
* Previous treatment with NB-UVB light or other light source within 6 weeks prior to the Screening Visit
* Patient not responsive to previous NB-UVB light treatment, defined as a patient who had undergone at least 20 NB-UVB sessions with no or minimal clinically relevant pigmentary response, in the opinion of the Investigator
* Previous topical treatment for vitiligo, including topical immunomodulators (e.g. corticosteroids, calcineurin inhibitors), within 4 weeks prior to the Screening Visit
* Allergy to afamelanotide or the polymer contained in the implant or to lignocaine/lidocaine or other local anaesthetic to be used during the administration of the implant
* History of photosensitivity disorders
* Claustrophobia
* Any active and/or unstable autoimmune disease judged to be clinically significant by the Investigator
* Any current skin disease that may have interfered with the study evaluation
* Female who was pregnant (confirmed by positive β-human chorionic gonadotropin (HCG) pregnancy test) or lactating
* Female of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives or diaphragm plus spermicide or intrauterine device) during the treatment phase (7 months) and for a period of three months thereafter - except if abstinence from intercourse was practiced
* Sexually active man with a partner of child-bearing potential (pre-menopausal, not surgically sterile) who was not using adequate contraceptive measures, as described above
* Participated in a clinical trial for an investigational agent within 30 days prior to the Screening Visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2016-02-02 (Actual); Study Completion 2016-06-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 participants were enrolled in the Arm Afamelanotide and NB-UVB (pooled analysis)
Groups:
- Afamelanotide and NB-UVB (Pooled Analysis): The study design was modified from a randomised controlled (Afamelanotide plus NB-UVB versus placebo plus NB-UVB) to an open label study (afamelanotide plus NB-UVB). A pooled analysis of all patients who received afamelanotide plus NB-UVB was undertaken and the results are presented.
Period: Overall Study
Arm/Group | Afamelanotide and NB-UVB (Pooled Analysis)
Started | 18
Completed | 15
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Afamelanotide and NB-UVB (Pooled Analysis)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Pigmentation (Total and Individual Body Parts) Using the Vitiligo Area Scoring Index (VASI)
Description: A decrease in VASI over time indicates a reduction of the body surface area affected by vitiligo and/ or a reduction in the body sites' degree of depigmentation (possible range 1-100)
Time Frame: From Day 0 to Day 196
Measure: Median (Full Range); unit: Change in VASI score from baseline
Arm/Group | Afamelanotide and NB-UVB (Pooled Analysis)
Number analyzed (Participants) | 15
Change in VASI score from baseline
  Total Day 28 | 0.00 [-0.63 to 0.25]
  Head and Neck Day 28 | 0.00 [-0.63 to 0.00]
  Hands Day 28 | 0.00 [0.00 to 0.00]
  Upper Extremities Day 28 | 0.00 [0.00 to 0.25]
  Trunk Day 28 | 0.00 [0.00 to 0.00]
  Lower Extremities Day 28 | 0.00 [0.00 to 0.00]
  Feet Day 28 | 0.00 [0.00 to 0.00]
  Total Day 56 | -0.05 [-2.25 to 1.00]
  Head and Neck Day 56 | 0.00 [-0.88 to 1.00]
  Hands Day 56 | 0.00 [-0.25 to 0.00]
  Upper Extremities Day 56 | 0.00 [-1.50 to 0.25]
  Trunk Day 56 | 0.00 [-1.00 to 0.00]
  Lower Extremities Day 56 | 0.00 [-2.25 to 0.00]
  Feet Day 56 | 0.00 [-0.20 to 0.00]
  Total Day 84 | -0.70 [-12.38 to 0.25]
  Head and neck Day 84 | 0.00 [-0.88 to 1.00]
  Hands Day 84 | 0.00 [-0.50 to 0.00]
  Upper Extremities Day 84 | 0.00 [-1.50 to 0.25]
  Trunk Day 84 | 0.00 [-7.75 to 0.00]
  Lower Extremities Day 84 | 0.00 [-4.50 to 0.00]
  Feet Day 84 | 0.00 [-0.20 to 0.00]
  Total Day 112 | -1.13 [-12.38 to 0.00]
  Head and Neck Day 112 | -0.10 [-1.00 to 0.50]
  Hands Day 112 | 0.00 [-0.50 to 0.00]
  Upper Extremities Day 112 | 0.00 [-3.00 to 0.25]
  Trunk Day 112 | -0.13 [-7.75 to 0.00]
  Lower Extremities Day 112 | 0.00 [-4.50 to 0.38]
  Feet Day 112 | 0.00 [-0.50 to 0.00]
  Total Day 140 | -2.56 [-15.15 to 0.00]
  Head and Neck Day 140 | -0.11 [-1.00 to 0.00]
  Hands Day 140 | 0.00 [-1.00 to 0.00]
  Upper Extremities Day 140 | -0.50 [-6.00 to 0.13]
  Trunk Day 140 | -0.50 [-7.75 to 0.00]
  Lower Extremities Day 140 | -0.50 [-5.85 to 0.38]
  Feet Day 140 | 0.00 [-0.50 to 0.00]
  Total Day 168 | -2.86 [-15.15 to 0.00]
  Head and Neck Day 168 | -0.13 [-1.00 to 0.00]
  Hands Day 168 | 0.00 [-1.00 to 0.00]
  Upper Extremities Day 168 | -0.50 [-6.00 to 1.00]
  Trunk Day 168 | -1.00 [-7.75 to 0.00]
  Lower Extremities Day 168 | -0.75 [-5.85 to 0.38]
  Feet Day 168 | 0.00 [-0.50 to 0.00]
  Total Day 196 | -3.70 [-15.65 to 1.00]
  Head and Neck Day 196 | -0.13 [-1.00 to 0.00]
  Hands Day 196 | 0.00 [-1.00 to 0.00]
  Upper Extremities Day 196 | -1.00 [-6.00 to 1.00]
  Trunk Day 196 | -1.13 [-7.75 to 0.75]
  Lower Extremities Day 196 | -0.60 [-5.85 to 0.38]
  Feet Day 196 | 0.00 [-0.50 to 0.00]

ADVERSE EVENTS:
Arm/Group | Afamelanotide and NB-UVB (Pooled Analysis)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide and NB-UVB (Pooled Analysis) (N=18)
Fatigue (General disorders) | 1
Glomerular filtration rate decreased (Investigations) | 1
Urinary casts (Investigations) | 1
Lethargy (Nervous system disorders) | 1
Nail pigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No